CLINICAL TRIAL: NCT04455009
Title: The Acute Effects of Fitness Drink Formulas Containing 100 mg and 140 mg of Caffeine on Energy Expenditure and Fat Metabolism in Healthy Adults
Brief Title: Acute Effects of Fitness Drink Formulas on Energy Expenditure and Fat Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Celsius Holdings, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BIO-17-13679
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Caffeine; Diet, Healthy; Fat Burn; Cognitive Change; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100mg Caffeine Formula (Experimental): 10kcal drink containing a total of 100 mg of caffeine from a proprietary blend of caffeine, guarana, ginger, and green tea extract containing epigallocatechin gallate
  Interventions: Dietary Supplement: Fitness Drink Formula
- 140mg Caffeine Formula (Experimental): 10kcal drink containing a total of 140 mg of caffeine from a proprietary blend of caffeine, guarana, ginger, and green tea extract containing epigallocatechin gallate
  Interventions: Dietary Supplement: Fitness Drink Formula
- Placebo Formula (Placebo Comparator): non-caloric/non-caffeinated drink
  Interventions: Dietary Supplement: Fitness Drink Formula

INTERVENTIONS:
Dietary Supplement: Fitness Drink Formula — Single drink provided following baseline assessments

SUMMARY:
The purpose of this investigation was to examine the acute effects of consuming two different fitness drink formulas on the physiological response at rest and to exercise in healthy men and women.

DETAILED DESCRIPTION:
Thermogenic fitness drinks containing ~200mg of caffeine have been reported to accelerate the metabolism, increase energy, and consequently promote increased fat oxidation. However, determination of the efficacy of lower caffeine concentrations may provide additional options for individuals with preferences for reduced caffeine intake. Therefore, the aim of this study was to evaluate different fitness drink formulas containing a total of 100mg and 140mg of caffeine on the physiological response at rest and to exercise.

This study utilized a randomized, double-blind, placebo-controlled design. All participants completed three testing visits during which they consumed the placebo, the 100mg caffeine formula, and the 140mg caffeine formula. Blood samples, blood pressure, heart rate, resting energy expenditure, substrate oxidation, and neurocognitive assessments were collected at baseline and repeated 30, 60, and 90 minutes post-ingestion. Immediately following the last cognitive assessment, a maximal graded exercise test with gas analysis was conducted on a cycle ergometer to evaluate physical performance and maximal fat oxidation during exercise as well as the physiological response prior to and following exercise.

ELIGIBILITY:
Inclusion Criteria:

* Young adult men and women between the ages of 18 and 35 years old.
* Participant is deemed by the investigator to be healthy and free of any physical limitations determined by physical activity readiness questionnaire (PAR-Q+) and medical and activity history questionnaire (MHQ).
* Participants will be required to be recreationally-active (defined according to American College of Sports Medicine standards of at least 150 minutes exercise per week and verified by information provided in the MHQ).
* Participant is willing to abstain from dietary supplementation throughout the duration of the study as indicated in the Informed Consent.
* Participant understands the study procedures and signs forms providing informed consent to participate in the study.

Exclusion Criteria:

* Inability to perform physical exercise, as determined by the PAR-Q+.
* Any "Yes" response in the PAR-Q+.
* History of hypertension, metabolic, hepatorenal, musculoskeletal, autoimmune or neurological disease, as determined by the MHQ.
* Regular consumption of greater than 250 mg per day of caffeine
* Currently taking thyroid, antihyperlipidemic, hypoglycemic, anti-hypertensive or androgenic medications.
* Taking any other nutritional supplement or performance-enhancing drug (determined from MHQ) that may interfere with the outcome variables of the study.
* Pregnancy (determined from MHQ).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Change in resting energy expenditure/substrate oxidation | Baseline, 30, 60, and 90 min post-ingestion
  Estimates from gas exchange analysis via indirect calorimetry
Change in energy expenditure/substrate oxidation in response to exercise | >90 min post-ingestion (pre/peri/post maximal graded exercise test)
  Estimates from gas exchange analysis via indirect calorimetry
Change in resting serum glycerol | Baseline, 30, 60, and 90 min post-ingestion
  Obtained from blood draw of the superficial forearm vein
Change in oxygen consumption/carbon dioxide production in response to exercise | >90 min post-ingestion (pre/peri/post maximal graded exercise test)
  Estimates from gas exchange analysis via indirect calorimetry
Change in resting minute ventilation | Baseline, 30, 60, and 90 min post-ingestion
  Estimates from gas exchange analysis via indirect calorimetry
Change in minute ventilation in response to exercise | >90 min post-ingestion (pre/peri/post maximal graded exercise test)
  Estimates from gas exchange analysis via indirect calorimetry

SECONDARY OUTCOMES:
Change in Automated Neuropsychological Assessment Metrics (ANAM) screening | Baseline, 30, 60, and 90 min post-ingestion
  Measures from mood scale, go/no go test, Stroop test
Change in resting blood pressure response | Baseline, 30, 60, and 90 min post-ingestion
  Measured via automated blood pressure monitor
Change in resting heart rate/heart rate variability | Baseline, 30, 60, and 90 min post-ingestion
  Measured via chest-based heart rate monitor
Change in heart rate/heart rate variability in response to exercise | >90 min post-ingestion (pre/peri/post maximal graded exercise test)
  Measured via chest-based heart rate monitor
Change in power output | >90 min post-ingestion
  Obtained via cycle ergometer during the maximal graded exercise test

CONTACTS AND LOCATIONS:
Overall Officials: David Fukuda, PhD, Principal Investigator — University of Central Florida
Locations (1):
- Kinesiology Laboratories, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No